CLINICAL TRIAL: NCT00362635
Title: A Double-blinded and Randomised Study to Compare the Efficacy and Safety of 48-week Treatment With Clevudine 30 mg qd Versus Lamivudine 100 mg qd for Chronic Hepatitis B Infection
Brief Title: Compare the Efficacy and Safety of 48-week Treatment With Clevudine 30mg Versus Lamivudine 100mg for CHB Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bukwang Pharmaceutical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLV-310
Record Dates: First submitted 2006-08-08; First posted 2006-08-10 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2012-07

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — clevudine

INTERVENTIONS:
Drug: Clevudine

SUMMARY:
The purpose of this study is to compare the efficacy and safety of 48-week treatment with Clevudine 30 mg qd versus lamivudine 100 mg qd for chronic hepatitis B infection.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is between 18 and 60, inclusive.
2. Patient is HBV DNA positive with DNA levels at screening >= 3 x 1,000,000 copies/mL.
3. Patient is documented to be HBsAg positive for > 6 months and HBeAg positive.
4. Patient has AST and ALT levels which are >= 1 times and <= 10 times the upper limit of normal (x ULN).
5. Patient has bilirubin levels <= 1.5 x ULN or bilirubin levels > 1.5 x ULN with diagnosis of Gilbert's disease and conjugated bilirubin within normal limits.
6. Women of childbearing age must have a negative urine (b-HCG) pregnancy test before start of trial treatment.
7. Patient is able to give written informed consent prior to study start and to comply with the study requirements.

Exclusion Criteria:

1. Patient is currently receiving antiviral, immunomodulatory or corticosteroid therapy.
2. Patients previously treated with lamivudine, lobucavir, adefovir, famciclovir, or any other investigational nucleoside for HBV infection.
3. Previous treatment with interferon must have ended at least 6 months prior to the screening visit.
4. Patient has a history of ascites, variceal hemorrhage or hepatic encephalopathy.
5. Patient is co-infected with HCV or HIV.
6. Patient has evidence of decompensated cirrhosis or hepatocellular carcinoma (alpha fetoprotein).
7. Patient is pregnant or breast-feeding.
8. Patient is unwilling to use an "effective" method of contraception during the study and for up to 3 months after the use of study drug ceases. For males, condoms should be used. Females must be surgically sterile (via hysterectomy or bilateral tubal ligation), post-menopausal, or using at least a medically acceptable barrier method of contraception (i.e., IUD, barrier methods with spermicide or abstinence).
9. Patient has a clinically relevant history of abuse of alcohol or drugs.
10. Patient has a significant gastrointestinal, renal, hepatic (decompensated), bronchopulmonary, neurological, cardiovascular, oncologic or allergic disease.
11. Subjects who are currently participating in another investigational study or has been taking any investigational drug within the last 4 weeks prior to Screening Visit.
12. Subjects who are taking any traditional Chinese medication, or has been taking any traditional Chinese medication within the last 2 weeks prior to Screening Visit.
13. Any criteria, which, in the opinion of the investigator, suggests that the subject would not be compliant with the study protocol.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Estimated)
Dates: Start 2006-08; Primary Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Efficacy: incident rate of the HBV DNA negativity (i.e. <300 copies/ml) by PCR
Safety: Laboratory tests, Adverse Events, Physical examination

SECONDARY OUTCOMES:
Efficacy:
Viral kinetics of HBV DNA suppression
Viral dynamic study over the first 12 weeks to define the nature of the anti-viral effect of Clevudine compared to Lamivudine.
Evaluation of the changes of ALT normalization rate and HBV serology over 48 weeks of treatment period
Evaluation of the proportion of patients with HBV DNA <300 copies/ml, median HBV DNA change from baseline(log10 copies/ml), the proportion of patients with normal ALT, and HBV serology over an additional 48 weeks of open label treatment

CONTACTS AND LOCATIONS:
Overall Officials: George KK Lau, M.D., Principal Investigator — Queen Mary Hospital, Hong Kong; Nancy Leung, M.D., Principal Investigator — Alice Ho Miu Ling Nethersole Hospital
Locations (2):
- Hong Kong (2):
  - Alice Ho Miu Ling Nethersole Hospital, Tai Po, New Territories
  - Queen Mary Hospital, Road

REFERENCES:
- See also: Unique trial number : HKCTR-250 — http://www.hkclinicaltrials.com/